CLINICAL TRIAL: NCT04963946
Title: STop and Restart Acalabrutinib In fRail Patients With Previously Untreated Chronic Lymphocytic Leukemia. A FILO Study.
Brief Title: STop and Restart Acalabrutinib In fRail Patients With Previously Untreated Chronic Lymphocytic Leukemia
Acronym: STAIR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FILOCLL14 - STAIR
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Untreated Chronic Lymphocytic Leukemia

STUDY DESIGN:
Intervention Model Description: multicenter, non comparative, randomized, stop and restart
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- watch and monitor (Experimental): After 18 months of acalabrutinib treatment, patients will stop acalabrutinib treatment for watch and monitor until month 60. If progression disease, patients will be re-treated with ACA at the last received dose after central reviewing of treatment criteria.
  Interventions: Drug: Stop ACA
- Acalabrutinib (Active Comparator): After 18 months of acalabrutinib treatment, patients will continue acalabrutinib treatment until month 60. If progression disease or unacceptable toxicity, patients will receive next line therapy at the discretion of their physicians and according to iwCLL 2018 criteria
  Interventions: Drug: ACA Continuation

INTERVENTIONS:
Drug: Stop ACA — discontinuation of acalabrutinib after 18 months in treatment-naïve CLL patients
  Arms: watch and monitor
Drug: ACA Continuation — continuation of acalabrutinib at the same dose
  Arms: Acalabrutinib

SUMMARY:
The irreversible Bruton's Tyrosine Kinase (BTK) inhibitor acalabrutinib (ACA) has potent clinical activity as a single agent in patients with treatment naive and Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL).

However, a growing body of concerns is raising regarding the unlimited administration of targeted therapy as BTKi. First, long-term treatments expose the patients to increased risk of specific adverse events (infections, bleeding events or cardiovascular problems). Second, continuous administration might also increase the risk of clonal evolution and therapeutic resistance resulting from genetic alterations such as BTK or PLCG2 mutations. Discontinuation of therapy after a fixed period is expected to prevent these events.

Rapid and deep responses yielded by ACA in elderly patients pave the way of investigating a limited 18-months period schedule. This study aims to investigate the 1-year PFS upon ACA discontinuation and efficacy of restarting ACA upon symptomatic relapse.

DETAILED DESCRIPTION:
This multicenter, non comparative, randomized phase II trial aims at evaluating the impact of a stopping ACA strategy on PFS of CLL patients >70 years or with coexisting comorbidities.

Patients will receive continuous Acalabrutinib (ACA) at 100 mg bid for 18 months. Dose adaptations will be made according to labels.

In case of first occurrence of grade ≥3 non-hematological toxicity, febrile grade ≥3 neutropenia or grade ≥4 hematological toxicity treatment must be stopped until recovering grade 1 or baseline state.

* 1st and second occurrence : restart at 100 mg twice daily
* 3rd occurrence : restart at 100 mg once daily
* 4th occurrence : discontinue acalabrutinib

At month 19 day 1, patients will be randomized (1:2) in two arms:

* Arm 1 = Control arm (acalabrutinib) continuing acalabrutinib until disease progression or unacceptable toxicity or
* Arm 2 = Experimental arm (watch and monitor) without ACA (see trial design).

Upon progression in the experimental arm, all patients will be re-treated with ACA at the last received dose after central reviewing of treatment criteria.

Upon progression in the control arm, patients will receive next line therapy at the discretion of their physicians and according to iwCLL 2018 criteria.

Patients will be monitored every three months until M31 then every 6 months until M60 or progression for both response and toxicity according to CTCAE v.5.

Minimal/Measurable Residual Disease (MRD) assessment will be done at month 19 day 1 in the peripheral blood.

CT-scan will be performed at baseline, then at month 19 day 1 and every 6 months within the year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Previously untreated CLL or Small Lymphocytic Lymphoma (SLL)
* CLL or SLL requiring treatment according to the iwCLL 2018 criteria2
* Total Cumulative Illness Rating Scale (CIRS) score > 6 or 30 < CrCl < 69 mL/min
* Both patients with or without TP53 disruption 17p deletion and/or TP53 mutations) can be included
* Patients can be included whatever their IGHV mutational status
* Patients with therapy-controlled cardiovascular comorbidities and/or anticoagulation (novel oral anticoagulant alone, aspirin alone, heparin alone) can be included (patients treated by vitamin K antagonist or dual anti-platelet therapy cannot be included)
* Life expectancy > 6 months
* Adequate hematology values: absolute neutrophil count ≥ 0.75 x 109/L, platelet count ≥ 50 x 109/L.
* Adequate liver function as indicated by a total bilirubin <1.5, aspartate transaminase and alanine transaminase ≤3 the institutional upper limits of normal values, unless directly attributable to CLL
* Signed (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including specify biology analysis, and are willing to participate in the study.

Exclusion Criteria:

* Known HIV seropositivity
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Known history of human immunodeficiency virus, serologic status reflecting active hepatitis B virus or hepatitis C virus infection, any uncontrolled active systemic infection along with subjects who are on ongoing anti-infective treatment and subjects who have received vaccination with a live attenuated vaccine within 4 weeks before the first dose of study treatment

    1. Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antibody (anti-HBs) negative will need to have a negative hepatitis B virus Polymerase Chain Reaction (PCR) result before enrollment. Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B virus PCR positive will be excluded.
    2. Subjects who are hepatitis C virus antibody positive will need to have a negative hepatitis C virus PCR result before enrollment. Those who are hepatitis C virus PCR positive will be excluded
  * Active and uncontrolled autoimmune cytopenia, including autoimmune hemolytic anemia (AIHA) (isolated positive Direct Antiglobulin Testing (DAT) is not an exclusion criteria) and idiopathic thrombocytopenic purpura (ITP).
  * Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura.
* Patients treated by vitamin K antagonist or dual anti-platelet therapy
* History of bleeding diathesis (e.g. hemophilia or von Willebrand disease)
* History of confirmed progressive multifocal leukoencephalopathy (PML).
* Concurrent severe diseases which exclude the administration of therapy :

  * heart insufficiency New York Heart Association (NYHA) grade III/IV, Left Ventricular Ejection Fraction (LEVF) < 50% and or Recirculation Fraction (RF) < 30%, myocardial infarction within the past 6 months prior to study
  * Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional (Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study)
  * severe chronic obstructive lung disease with hypoxemia
  * history of stroke or intra-cranial hemorrhage within the last 6 months
  * severe diabetes mellitus
  * uncontrolled hypertension
  * impaired renal function with creatinine clearance < 30 ml/min according the formula of Cockcroft and Gault
  * Patient who requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment in this study.
* Disease significantly affecting gastrointestinal function (malabsorption syndrome, stomach or small bowel resection)
* Evidence for Richter syndrome
* Treatment with any of the following within 7 days prior to the first dose of study drug: steroid therapy for anti-neoplastic intent.
* A significant history of renal, neurologic, psychiatric, endocrine, metabolic, immunologic, cardiovascular, or hepatic disease that, in the opinion of the investigator, would adversely affect the patient's participation in this study or interpretation of study outcomes
* Major surgery within 30 days prior to the first dose of study treatment.
* History of prior other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following:

  * curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study.
  * other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which patient is disease-free for ≥ 5 years without further treatment
* Adult under law-control
* Fertile male patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study
* No affiliation to social security

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at one year after acalabrutinib interruption | until 12 months after acalabrutinib interruption
  Time from randomization (M19 : discontinuation of acalabrutinib after of 18 months treatment) to progression (needing therapy or not) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Ysebaert, Pr, Principal Investigator — French Innovative Leukemia Organisation; Romain GUIEZE, Pr, Principal Investigator — French Innovative Leukemia Organisation
Locations (32):
- France (32):
  - Chu Angers, Angers
  - ARGENTEUIL - Centre hospitalier Victor Dupouy, Argenteuil
  - Ch Avignon, Avignon
  - Ch Cote Basque, Bayonne
  - BOBIGNY - Hôpital Avicenne, Bobigny
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - Corbeil-Essonnes -, Corbeil-Essonnes
  - CHU Grenoble - Hématologie, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Léon Bérard - Hématologie, Lyon
  - Institut Paoli-Calmettes - Hématologie Clinique, Marseille
  - Centre Hospitalier Regional Metz Thionville, Metz
  - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - Hopital E.Muller, Mulhouse
  - CHR ORLEANS - Hématologie, Orléans
  - Hopital Pitie Salpetriere Service Hematologie Clinique - Pavillon de L'Enfant Et Adolescent, Paris
  - CENTRE HOSPITALIER SAINTJEAN - Hématologie Clinique, Perpignan
  - Bordeaux Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie - Hématologie et Thérapie Cellulaire, Poitiers
  - CERGY-PONTOISE - Centre Hospitalier René Dubos, Pontoise
  - Chu Reims, Reims
  - CHU Pontchaillou - Hématologie Clinique BMT-HC, Rennes
  - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - IUCT ONCOPOLE - Hématologie, Toulouse
  - Hôpital Bretonneau - Hématologie et Thérapie Cellulaire, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Vannes - Chba, Vannes
  - VERSAILLES - Hôpital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: No